CLINICAL TRIAL: NCT02195271
Title: Effect of Melatonin and Transcranial Direct Current Stimulation (tDCS) on Neuroplasticity and the Heat-pain Detection Threshold in Healthy Subjects:Randomized, Double-blind,Crossover Trial
Brief Title: Neuroplasticity:Melatonin and Transcranial Current Stimulation in Healthy Subjects.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 130155
Record Dates: First submitted 2014-03-19; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Analgesia Disorder; Pain
Keywords: Melatonin; Transcranial Direct Current Stimulation; Neuroplasticity; Analgesia; Pain
MeSH Terms: conditions — Pain; Agnosia | interventions — Transcranial Direct Current Stimulation; Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Active Comparator): 0,25mg/Kg sl before tDCS
  Interventions: Drug: Melatonin
- tDCS (Experimental): Transcranial direct current stimulation once time. Dose 2 mA, 20 seconds.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS)
  Arms: tDCS
Drug: Melatonin
  Arms: Melatonin

SUMMARY:
Pain exerts a tremendous cost in healthy care, rehabilitation and lost productivity. It is is associated with a wide range of diseases and their social consequences is a public health problem.

With the progress of neuroscience and studies on the plasticity of the central nervous system, it has been provided a better understanding of the neurobiological mechanisms of pain.

The neurohormone Melatonin stands by having systemic and diverse mechanisms of action, both in physiological and pathological situations, with modulating effects on the process of nociceptive signaling and neurochemical mechanisms such as serotonergic, opioidergic and GABAergic, exerting anti-inflammatory action, analgesic activity among others.

The advent of neuromodulation techniques such as transcranial direct current stimulation (tDCS), which promote changes in neuronal activity and signaling to be effective in conditions of chronic pain by attenuating changes in cortical excitability.

There is clinical evidence of the analgesic effect of Melatonin and tDCS alone. Thus, considering the potential for each isolated intervention and the lack of knowledge of their combined effect, the authors propose the present study to investigate the effect of this combination on the heat-pain detection threshold and the neuroplasticity in the healthy subjects.

DETAILED DESCRIPTION:
The methods are according to the CONSORT guidelines.

Heat pain threshold and tolerance : Quantitative Sensory Testing (QST) will be used on a computer Peltier-based device thermode.

Conditioned Pain Modulation (CPM)-task: Immerssing the non-dominant hand cold water for 1 minute.

Serum Brain Derived Neurotrophic Factor (BDNF).

Transcranial Magnetic Stimulation (TMS) assessment: motor threshold, motor evoked potential, Short intracortical inhibition and intracortical facilitation.

Statistical analyses: Descriptive statistics, Linear and multiple regression analysis, performed with SPSS version18.0.

ELIGIBILITY:
Inclusion Criteria:

* Male 18-40 years old
* Healthy
* Without medication
* Sign the informed consent

Exclusion Criteria:

* Patients who did not understand the Portuguese
* Acute or chronic pain conditions
* Medical or psychiatric disorders
* History of alcohol or substance abuse
* Neurological disorder
* Use of medications affect in the central nervous system
* Traumatic brain injury
* Neurosurgery
* Metallic implant in the brain

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in heat-pain threshold with pain score | Baseline, one week
  Heat-threshold by Pettier-based device on the contralateral hand assessment pain score (VAS)

SECONDARY OUTCOMES:
Change from baseline Brain-Derived neurotrophic factor (BDNF) | Baseline, one week
Change from Baseline from Catastrophizing Scale | Baseline, one week
Change from baseline Inventory of state-trait anxiety Scale | Baseline, one week
Change from baseline Inventory of Coping | Baseline, one week
Change from baseline of cortical excitability | Baseline, one week
  Transcranial Magnetic Stimulation (TMS) assessment motor threshold, motor-evoked potentials, silent period, intracortical inhibition and facilitation

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, Principal Investigator — Hospital de Clinicas de Porto Alegre - UFRGS
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil